CLINICAL TRIAL: NCT01217359
Title: Differences in Evoked Intracellular Interferon Signaling Pathways Using Single Cell Phosphoprotein Profiling
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 08-2040
Record Dates: First submitted 2010-09-30; First posted 2010-10-08 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Interferon alpha-2; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interferon Alfa-2b (Experimental): Patients will receive a single dose of interferon
  Interventions: Drug: Interferon Alfa-2b

INTERVENTIONS:
Drug: Interferon Alfa-2b — Patients will receive a single dose of interferon followed by serial blood draws to assess cellular responses to interferon
  Other Names: Intron A

SUMMARY:
Purpose:

The purpose of this exploratory study is to evaluate phosphoprotein profiling to determine differences in the intracellular actions of interferon or interferon stimulated genes among people with different treatment outcomes to interferon based therapy for hepatitis C (HCV). Participants: Patients with genotype 1 HCV who have had interferon based therapy at the University of North Carolina (UNC). Procedures: Thirty patients with varied responses to treatment will be given a single subcutaneous injection of interferon alpha 2b. Prior to the injection and at 30 minutes, 1,2,4,6,12 and 20 hours after injection, blood will be drawn for analysis of phosphoprotein profiling and changes in serum cytokines.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, subjects must meet the following inclusion criteria:

* Willing and able to provide informed consent
* Males or females age 18 - 65 years
* For women of childbearing potential, negative blood pregnancy test documented within the 24-hour period prior to IFN-α administration
* History of genotype 1 HCV infection previously treated with peginterferon and ribavirin and with a virological response that can be determined from retrospective review of medical records
* A washout period of >12 weeks between the last dose of prescribed peginterferon and ribavirin and the screening visit

Exclusion Criteria

Subjects with any of the following will not be eligible for participation:

* Neutrophil count <1500 cells/mm3, Hgb <12 g/dL in women or 13 g/dL in men, or platelet count <75,000 cells/mm3 at screening
* Serum creatinine level >1.5 times the upper limit of normal at screening
* Poorly controlled psychiatric illness, as determined by the study physician, which can be exacerbated by interferon therapy
* Infection requiring antibiotics, symptomatic viral infection, inflammatory process requiring therapy, or allergic reactions in the week immediately preceding the inpatient study visit
* Use of medications that affect the immune system (e.g. glucocorticoids, chronic NSAIDs daily) in the week immediately preceding the inpatient study visit
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, psoriasis, rheumatoid arthritis)
* Women with ongoing pregnancy or breast-feeding
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* History of a seizure disorder or current anticonvulsant use
* History of major organ transplantation with an existing functional graft
* History of thyroid disease poorly controlled on prescribed medications
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Protein quantification of interferon stimulated genes (ISG) | 0-20 hours
  This is an exploratory study observing downstream phosphorylation of interferon stimulated genes in the Janus Activated Kinase (JAK-STAT) pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Sid Barritt, MD, MSCR, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No